CLINICAL TRIAL: NCT01420406
Title: Impact of Daily Feeding of Food Sources of Cryptoxanthin (CX) and Beta-carotene (BC) on Plasma and Breast Milk Concentrations of CX, BC, and Retinol (VA) in Lactating Women With Marginal Vitamin A Status
Brief Title: Vitamin A Bioavailability in Lactating Women With Marginal Vitamin A Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: WHNRC 200816672
Record Dates: First submitted 2011-08-17; First posted 2011-08-19 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Vitamin A Deficiency
Keywords: lactation; cryptoxanthin; beta-carotene; vitamin A
MeSH Terms: conditions — Vitamin A Deficiency; Breast Feeding

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 0 mg retinol (Placebo Comparator): 0 mg retinol activity equivalents (RAE) as white-fleshed sweet potatoes and a corn oil capsule
  Interventions: Other: 0 mg retinol activity equivalents
- 12 mg BC (Experimental): 12 mg of BC as orange-fleshed sweet potatoes and a corn oil capsule.
  Interventions: Other: 12 mg of BC
- 6 mg of CX (Experimental): 6 mg of CX as tangerines and a corn oil capsule
  Interventions: Other: 6 mg of CX
- 1.0 mg RAE (Experimental): 1.0 mg RAE vitamin A as retinyl palmitate in corn oil, and white-fleshed sweet potatoes
  Interventions: Other: 1.0 mg RAE

INTERVENTIONS:
Other: 0 mg retinol activity equivalents — 0 mg retinol activity equivalents (RAE) as white-fleshed sweet potatoes and a corn oil capsule
  Arms: 0 mg retinol
Other: 12 mg of BC — 12 mg of BC as orange-fleshed sweet potatoes and a corn oil capsule
  Arms: 12 mg BC
Other: 6 mg of CX — 6 mg of CX as tangerines and a corn oil capsule
  Arms: 6 mg of CX
Other: 1.0 mg RAE — 1.0 mg RAE vitamin A as retinyl palmitate in corn oil, and white-fleshed sweet potatoes
  Arms: 1.0 mg RAE

SUMMARY:
The study will assess the relative bioavailability and bioefficacy of cryptoxanthin (CX) and beta-carotene (BC) from food sources for increasing breast milk carotenoid and retinol concentrations in lactating Bangladeshi women.

DETAILED DESCRIPTION:
The specific aim is to compare the effects of orange-fleshed sweet potatoes and tangerines compared to white-fleshed sweet potatoes and vitamin A as retinyl palmitate on blood and breast milk cryptoxanthin (CX), beta-carotene (BC), and vitamin A (VA) concentrations by randomly assigning lactating Bangladeshi women to one of four treatment groups for 6 days/week for 3 weeks.

The investigators will also compare the relative vitamin A (VA) value of BC and CX from food sources by comparing the mean change in breast milk retinol concentrations of the groups that receive tangerines (CX) or orange-fleshed sweet potatoes (BC) with the mean change in breast milk retinol of the group that receives retinyl palmitate.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women in Dhaka, Bangladesh
* Lactating women in their 2nd or 3rd month of lactation who are planning to breast-feed at least 6 months
* Breast-feeding only one infant
* Age range 18 to 45 years
* Not pregnant
* Serum retinol concentrations >0.70 umol/L and <1.10 umol/L
* Normal concentrations of CRP (<10 mg/L)
* At least one arm vein deemed adequate for blood collection, as evaluated by a screening nurse.
* Willing to consume the test foods daily 6 d/wk for one month

Exclusion Criteria:

* Health status is not compatible with the inclusion criteria, such as screening blood chemistries indicative of vitamin A deficiency.
* Severe anemia (Hb <9 mg/dL)
* Current pregnancy
* Must not have known allergy to citrus fruit (tangerines or mandarin oranges) or sweet potatoes
* Must have no obvious psychological or sociological problems-such as alcoholism, drug abuse, or severe and acute mental illness that would influence their ability to sign an inform consent agreement or to participate in study duties and activities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2010-06; Primary Completion 2011-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change in carotenoids in serum and breast milk | 1 and 3 weeks
  We will measure serum and breast milk beta-carotene, beta-cryptoxanthin, other carotenoids, and vitamins A and E.

SECONDARY OUTCOMES:
Change in Dark adaptation | 1 and 3 weeks
  Dark adaptation will be measured by the pupillary threshold (PT) test on the first and 3rd weeks of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Betty J Burri, PhD, Principal Investigator — WHNRC
Locations (1):
- International Centre for Diarrhoeal Disease Research, Dhaka, Bangladesh

REFERENCES:
- [Derived] Turner T, Burri BJ, Jamil KM, Jamil M. The effects of daily consumption of beta-cryptoxanthin-rich tangerines and beta-carotene-rich sweet potatoes on vitamin A and carotenoid concentrations in plasma and breast milk of Bangladeshi women with low vitamin A status in a randomized controlled trial. Am J Clin Nutr. 2013 Nov;98(5):1200-8. doi: 10.3945/ajcn.113.058180. Epub 2013 Sep 4. PMID 24004891